CLINICAL TRIAL: NCT00446706
Title: Estimation of Intrinsic Positive End-Expiratory Pressure (PEEP) in Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Juan B. Figueroa-Casas, Associate Professor, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: Estimation PEEPi
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Intrinsic PEEP
MeSH Terms: conditions — Respiratory Distress Syndrome; Positive-Pressure Respiration, Intrinsic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
ARDS (Acute Respiratory Distress Syndrome) is a condition of severe inflammation and excess fluids in the lungs that impairs their function of oxygen uptake to the point of needing a ventilator (breathing machine) to help them obtain enough oxygen into the body. Because of the high amounts of gas that the ventilator has to give to these patients, high pressures may develop deep into the lungs and produce complications for the patient. However, physicians sometimes cannot recognize it because it requires special equipment to measure pressure deep in the lungs. The goal of this study is to determine if the amount of this pressure can be calculated using mathematical formulas and the routine numbers provided by ventilators. The study consists on making the conventional measurement of this deep pressure and at the same time calculate this same pressure from other measurements that the ventilator routinely provides, to see if the calculated value can replace the more complicated conventional measurement. The measurements will be done by:

1. placing a small device along the tubing connecting the patient to the ventilator;
2. giving medicines to relax the muscles (if the patient is not already receiving them); and
3. making the ventilator hold the patient's breath for a few seconds to take measurements.

This is repeated after the breathing rate of the ventilator is increased or decreased mildly. Risks related to the medicine to be used and the measuring maneuvers are rare but include transient narrowing of windpipes, transiently low heart rate, blood pressure or blood oxygen, and allergic reactions. This is not a treatment. The information obtained during the study will be shared with the treating doctors who may find it useful to make adjustments to the ventilator. The patient may receive no direct benefit from being in this study; however, the findings may contribute to better care for this kind of patients in the future.

DETAILED DESCRIPTION:
Intrinsic PEEP (Positive-End Expiratory Pressure) was measured by end-expiratory occlusion method and estimated using formulas derived from measured expiratory flows and a postulated linear pressure-flow relationship during expiration in passive ARDS patients. Agreement between measured and estimated intrinsic PEEP was analyzed by Bland and Altman's method.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with diagnosis of ARDS, as defined by the American- European Consensus Conference 4
* Receiving mechanical ventilation.
* Presence of autoPEEP by inspection of flow-time waveforms displayed by the mechanical ventilator.

Exclusion Criteria:

* Known or suspected diagnosis of COPD or airflow limitation.
* Next of kin not available to consent.
* Contraindication to receive a muscle relaxant when measurements may be inaccurate without its administration.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Acute Respiratory Distress Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2004-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Agreement between Measured and Estimated Intrinsic PEEP | The day and time of measurement
  Bias and its standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Juan Figueroa-Casas, MD, Principal Investigator — Texas Tech University
Locations (1):
- Thomason Hospital (Now University Medical Center), El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No